CLINICAL TRIAL: NCT01604876
Title: Effect of Bright Light on Mood and Sleep in Parkinson's Disease
Acronym: LightPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: International Parkinson Foundation ('IPF'), Hoofddorp, The Netherlands (Unknown); Parkinsonvereniging, Bunnik, the Netherlands (Unknown); Netherlands Brain Foundation (Other); Netherlands Institute for Neurosciences, Amsterdam, The Netherlands (Unknown); GGZ inGeest (Other)
Responsible Party: Principal Investigator, O.A. van den Heuvel, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL3905802912
Record Dates: First submitted 2012-05-17; First posted 2012-05-24 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinson's disease; depression; light therapy; sleeping problems
MeSH Terms: conditions — Parkinson Disease; Depression; Parasomnias | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- light condition 1 + day night structure (Experimental): exposure to 10.000 lux light twice daily (morning + evening) for 30 minutes during 3 months at home.
  Interventions: Device: light therapy 30 min morning and evening, three months
- light condition 2 + day night structure (Active Comparator): exposure to 200 lux light twice daily (morning + evening) for 30 minutes during 3 months at home.
  Interventions: Device: light therapy 30 min morning and evening, three months

INTERVENTIONS:
Device: light therapy 30 min morning and evening, three months — Light from a commercially available table-mounted lightbox (Brazil, Lumie, Cambridge UK) [dimensions 50.2 x 32 x 15.4 cm] equipped with 3x36W Fluorescent bulbs (Osram 954), reflectors and a diffuser screen providing 10,000 lux at 30 cm eye level distance.
  therapy consists of 30 minutes light exposure in the morning and evening during 3 months.
  Other Names: light condition 1
  Arms: light condition 1 + day night structure
Device: light therapy 30 min morning and evening, three months — 200 lux light from a commercially available table-mounted lightbox (Brazil, Lumie, Cambridge UK) [dimensions 50.2 x 32 x 15.4 cm] To lower the intensity to 200 lux the bulbs are enwrapped with one layer of L299s neutral density filter (LEE Filters, Andover, UK).
  Therapy consists of 30 minutes light exposure in the morning and evening during 3 months.
  Other Names: light condition 2
  Arms: light condition 2 + day night structure

SUMMARY:
The purpose of this clinical trial is to investigate whether light therapy is a suitable treatment option for depression and insomnia in Parkinson's disease.

DETAILED DESCRIPTION:
The quality of life of patients with Parkinson's disease and their caretakers is mainly influenced by so called non-motor symptoms. This includes neuropsychiatric consequences of the disease like depression and sleeping problems. The incidence of depressed mood in patients with Parkinson is approximately 50%, the incidence for sleeping problems is 90%. These symptoms are often overlooked and even if recognized, inadequately treated. The treatment of mood and sleep disturbances in Parkinson patients is hampered by adverse effects, incomplete responses to the usual treatments and the absence of specific treatment options for these symptoms in Parkinson's disease. On the basis of the hypothesis of disturbed functioning of the suprachiasmatic nucleus in Parkinson's disease it is expected that stimulation of this nucleus by bright light therapy will result in improved functioning on multiple different domains: mood, sleep, motor functions, quality of life and circadian rhythms. Because there are virtually no side effects and the possibility of home treatment, light therapy is expected to be highly appreciated by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* depression

Exclusion Criteria:

* psychosis
* mania
* suicidality
* retinopathy
* previous light treatment
* use of photosensitising medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Mood | T0: baseline, T1: change from T0, T2: change from T0, T3: follow-up, change from T0, T4: follow-up, change from T0, T5: follow-up, change from T0
  using Hamilton Depression Rating Scale (HDRS - 17 items) and Geriatric Depression Scale-30 (GDS - 30 items) at baseline (T0), halfway therapy, six weeks (T1), end of therapy, three months (T2), at 1 month follow-up (T3), 3 months follow-up (T4) and 6 months follow-up (T5).
  * The direct treatment effect (= difference score between baseline and end of treatment),
  * The long-lasting treatment effect (= difference score between baseline and end of follow-up).
  * The dichotomous treatment response (> 50 % decrease score at T2), in order to calculate the Numbers Needed to Treat (NNT).

SECONDARY OUTCOMES:
Sleep | T0: baseline, T1: change from T0, T2: change from T0, T3: follow-up, change from T0, T4: follow-up, change from T0, T5: follow-up, change from T0
  using Scales for Outcomes in Parkinson's Disease-Sleep subscale (SCOPA-sleep - 14 items) assessed at baseline (T0), after 6 weeks of light therapy (T1), after 3 months of light therapy (end of treatment, T2), 1 month post-treatment (T3), 3 months post-treatment (T4) and 6 months post-treatment (T5).
Motor function | T0: baseline, T2: after three months therapy, change from T0, T5: six month follow-up, change from T0
  using Unified Parkinson's Disease Rating Scale-Section III motor score (UPDRS-III - 14 items) at 3 time points: at baseline (T0), after 3 months of light therapy (T2) and 6 months follow-up (T5).
Quality of Life of patient | T0: baseline, T2: after three months therapy, change from T0, T5: six month follow-up, change from T0
  using the World Health Organization Quality of Life Assessment Short Version (WHOQOL-BREF) assessed at 3 time points, at baseline (T0), after 3 months of light therapy (T2) and 6 months follow-up (T5).
Circadian rhythm | T0: baseline, T1: change from T0, T2: change from T0, T3: follow-up, change from T0, T4: follow-up, change from T0, T5: follow-up, change from T0
  Circadian rhythm as measured by melatonin and cortisol day/night curves and actigraphy are assessed at 6 time points, at baseline (T0), after 6 weeks of light therapy (T1), after 3 months of light therapy (T2), 1 month follow-up (T3), 3 months follow-up (T4) and 6 months follow-up (T5).
Quality of life of caregiver | T0: baseline, T2: after three months therapy, change from T0, T5: six month follow-up, change from T0
  using the Zarit Burden Interview (ZBI - 22 items) for caregivers, assessed at 3 time points, at baseline (T0), after 3 months of light therapy (T2) and 6 months follow-up (T5).

CONTACTS AND LOCATIONS:
Overall Officials: Odile A van den Heuvel, MD PHD, Principal Investigator — Amsterdam UMC, location VUmc; Ysbrand D van der Werf, PHD, Principal Investigator — Amsterdam UMC, location VUmc; Jan H Smit, PHD, Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared on reasonable request

REFERENCES:
- [Derived] Rutten S, Vriend C, Smit JH, Berendse HW, van Someren EJW, Hoogendoorn AW, Twisk JWR, van der Werf YD, van den Heuvel OA. Bright light therapy for depression in Parkinson disease: A randomized controlled trial. Neurology. 2019 Mar 12;92(11):e1145-e1156. doi: 10.1212/WNL.0000000000007090. Epub 2019 Feb 15. PMID 30770426
- [Derived] Rutten S, Vriend C, Smit JH, Berendse HW, Hoogendoorn AW, van den Heuvel OA, van der Werf YD. A double-blind randomized controlled trial to assess the effect of bright light therapy on depression in patients with Parkinson's disease. BMC Psychiatry. 2016 Oct 21;16(1):355. doi: 10.1186/s12888-016-1050-z. PMID 27769202